CLINICAL TRIAL: NCT02710994
Title: A Randomized, Open Label, Two-way Crossover Designed Clinical Trial to Investigate the Pharmacodynamics and the Safety Between Repeated Doses of CDFR0209 in Healthy Male Volunteers
Brief Title: Pharmacodynamics and Safety of CDFR0209
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: CTC Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED-CT1-14-085
Record Dates: First submitted 2016-03-04; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Stomach Ulcer; Gastroesophageal Reflux
Keywords: Immediate release omeprazole; Integrated gastric acidity
MeSH Terms: conditions — Stomach Ulcer; Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDFR0209, Then Losec (Experimental): Subjects first received CDFR0209 each morning in a fasting state for 7 days. After a washout period of 14 days, they then received Losec 40 mg in a fasting state each morning for 7 days.
  Interventions: Drug: CDFR0209; Drug: Losec
- Losec, Then CDFR0209 (Experimental): Subjects first received Losec 40 mg each morning in a fasting state for 7 days. After a washout period of 14 days, they then received CDFR0209 in a fasting state each morning for 7 days.
  Interventions: Drug: CDFR0209; Drug: Losec

INTERVENTIONS:
Drug: CDFR0209 — Immediate release omeprazole 40 mg and sodium bicarbonate 1,100 mg
Drug: Losec — Losec 40 mg

SUMMARY:
This is a randomized, open-label, two-way crossover study to investigate the pharmacodynamics(24 hour gastric pH) and the safety between repeated doses of CDFR0209 and Losec in Healthy Male Volunteers

DETAILED DESCRIPTION:
Eligibility for participation of this study was determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study were admitted to the Clinical Trial Center of Ajou University Medical Center on the 2 day before dosing (Day -2).

On Day -1 around 8 AM, ambulatory intragastric pH recording was performed using ZepHr® pH Monitoring System (Sandhill Scientific, Inc., Highlands Ranch, CO, USA) without dosing for 24 hours.

On Day 1, subjects was dosed Losec 40 mg or CDFR0209 (Omeprazole 40 mg & sodium bicarbonate 1,100 mg) around 8 AM and ambulatory intragastric pH recording was continued upto 24 hours after dosing.

From Day 2 ~ 6, subjects were dosed Losec 40 mg or CDFR0209 around 8 AM. On Day 7, subjects was dosed Losec 40 mg or CDFR0209 (Omeprazole 40 mg & sodium bicarbonate 1,100 mg) around 8 AM and ambulatory intragastric pH recording was performed upto 24 hours after dosing.

After 14 days of washout period, subjects was dosed Losec 40 mg or CDFR0209 by crossover manner and ambulatory intragastric pH recording was performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* With in 20% of ideal body weight, {Ideal body weight=[height(cm)-100]*0.9}
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal disease or mental disorder (Past history or present)
* Inadequate result of laboratory test (especially, AST/ALT > 1.25 x UNL, Total bilirubin > 1.5 x UNL)
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL test and Helicobacter Ab IgM
* Positive result in urea breath test
* Taking OTC(Over the counter)medicine including oriental medicine within 7 days
* Clinically significant allergic disease (Except for mild allergic rhinitis and dermatitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to omeprazole and sodium bicarbonate
* Previous whole blood donation within 60 days or component blood donation within 30 days
* Previous participation of other trial within 90 days
* Continued taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean percent decrease from baseline in integrated gastric acidity after 7th dose | Day 7 upto 24 hours
  Data for 24 hour gastric pH were acquired at baseline (day -1) and day 7 of dosing with either Losec 40 mg or CDFR0209.
  Percent decrease from baseline in integrated gastric acidity after 7th dose = [Baseline integrated acidity - Day 7 integrated acidity]/ Baseline integrated acidity × 100.

SECONDARY OUTCOMES:
Mean percent decrease from baseline in integrated gastric acidity after 1st dose | Day 1 upto 24 hours
  Data for 24 hour gastric pH were acquired at baseline (day -1) and day 1 of dosing with either Losec 40 mg or CDFR0209.
  Percent decrease from baseline in integrated gastric acidity after 1st dose = [Baseline integrated acidity - Day 1 integrated acidity]/ Baseline integrated acidity × 100.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Medical Center, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No